CLINICAL TRIAL: NCT00314912
Title: An Open-Label Extension of the Phase III Study CL-758007 With Tramiprosate (3APS) in Patients With Alzheimer's Disease
Brief Title: Open-Label Extension of the Phase III Study With Tramiprosate (3APS) in Patients With Mild to Moderate Alzheimer's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-758017
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2007-07-16 (Estimated); Status verified 2007-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tramiprosate

INTERVENTIONS:
Drug: Tramiprosate (3APS)

SUMMARY:
The purpose of this Phase III open-label extension study is to evaluate the long-term safety of Tramiprosate (3APS) in patients with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
Duration of treatment: 12 months. Patients who complete the Phase III clinical trial will be offered the opportunity to receive Tramiprosate (3APS) in an open-label extension study

ELIGIBILITY:
Inclusion Criteria:

* The patient must have successfully completed the full 78-week duration of the double-blind CL-758007 study.
* Male or female (age 50 years and older): Female must be of non-childbearing potential (i.e. surgically sterilized or at least 2 years post-menopausal).
* Patient must be living in the community with a reliable caregiver. Participant living in an assisted living facility may be included if study medication intake is supervised and participant has a reliable caregiver.
* The patient must be presenting a reasonably good nutritional status.
* Signed inform consent from the patient or legal representative.

Exclusion Criteria:

Patients will not be eligible to participate in the study if they meet any of the following criteria:

* The patient participates in another drug trial during the study.
* The patient with a clinically significant and/or uncontrolled condition or other significant medical disease.
* The patient is unable to swallow medication tablets.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 2006-05

PRIMARY OUTCOMES:
To evaluate the long-term safety of Tramiprosate (3APS).

SECONDARY OUTCOMES:
To provide additional long-term data on the efficacy of Tramiprosate (3APS).

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Clinical Research Center, San Francisco, California, United States